CLINICAL TRIAL: NCT02716194
Title: A Phase 1, Prospective, Open Label, Two Period, Fixed Sequence, Dose-Escalation Study of the PK and Safety of BAX 826 (PSA-rFVIII) in Previously Treated Patients With Severe (FVIII <1%) Hemophilia A
Brief Title: BAX 826 Dose-Escalation Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 291501; 2015-004079-60 (EudraCT Number)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 - Low dose (Experimental): The study is comprised of 3 dose cohorts and two dose escalation steps [Cohort 1: 10 evaluable participants; Cohort 2: 10 evaluable participants; Cohort 3: 10 evaluable participants]. Participants will be recruited to the next dose level only after short-term safety has been reviewed and subject to approval by a Safety Review Committee at the preceding dose level.
  Interventions: Biological: BAX 826; Biological: Octocog alfa
- Cohort 2 - Medium dose (Experimental): The study is comprised of 3 dose cohorts and two dose escalation steps [Cohort 1: 10 evaluable participants; Cohort 2: 10 evaluable participants; Cohort 3: 10 evaluable participants]. Participants will be recruited to the next dose level only after short-term safety has been reviewed and subject to approval by a Safety Review Committee at the preceding dose level.
  Interventions: Biological: BAX 826; Biological: Octocog alfa
- Cohort 3 - High dose (Experimental): The study is comprised of 3 dose cohorts and two dose escalation steps [Cohort 1: 10 evaluable participants; Cohort 2: 10 evaluable participants; Cohort 3: 10 evaluable participants]. Participants will be recruited to the next dose level only after short-term safety has been reviewed and subject to approval by a Safety Review Committee at the preceding dose level.
  Interventions: Biological: BAX 826; Biological: Octocog alfa

INTERVENTIONS:
Biological: BAX 826
  Other Names: BAX826
Biological: Octocog alfa
  Other Names: ADVATE (Antihemophilic Factor [Recombinant]); ADVATE

SUMMARY:
1. To assess tolerability and safety of BAX 826 after a single infusion in previously treated patients (PTPs) with severe hemophilia A
2. To determine the pharmacokinetic (PK) parameters of BAX 826 compared to ADVATE
3. To evaluate immunogenicity of polysialic acid linked to Factor VIII (FVIII)

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated male participants aged 18 to 65 years (inclusive) at the time of screening
2. Diagnosis of severe hemophilia A (Factor VIII level <1%)
3. Previously treated with FVIII concentrates for ≥150 documented Exposure Days (EDs)
4. Karnofsky performance score of ≥60
5. Human immunodeficiency virus negative (HIV-); or HIV+ with stable disease
6. Hepatitis C virus negative (HCV-); or HCV+ with chronic stable hepatitis as assessed by the investigator
7. Able to understand and have provided written informed consent including signature on an informed consent form (ICF) approved by an ethics committee (EC)
8. Have provided written authorization for use and disclosure of protected health information
9. Agree to abide by the study schedule and to return for the required assessments
10. Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Detectable FVIII inhibitor at screening, with a titer ≥0.6 Bethesda Unit (BU)
2. Documented history of FVIII inhibitors with a titer ≥0.4 BU at any time prior to screening
3. Known clinical hypersensitivity towards mouse or hamster proteins or to polysialic acid (PSA)
4. Scheduled elective surgery during study participation
5. Severe chronic hepatic dysfunction
6. Severe renal impairment
7. Currently receiving, or has recently received (less than 3 months prior to study participation), or is scheduled to receive during the course of the study, other PSA-ylated drugs
8. Have received another investigational drug within 30 days prior to study entry and/or is scheduled to receive additional investigational drug during the course of the study in the context of another investigational drug study
9. Diagnosis of an inherited or acquired hemostatic defect other than hemophilia A
10. Currently receiving, or scheduled to receive during the course of the study, an immune-modulating drug other than antiretroviral chemotherapy
11. Has a clinically significant medical, psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the investigator, would affect the safety or compliance of the participant during the study
12. Is a family member or employee of the investigator

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (28):
- UMHAT "Sv. Georgi", EAD, Plovdiv, Bulgaria
- Germany (5):
  - Werlhof-Institut, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Vivantes Klinikum im Friedrichshain - Landsberger Allee, Berlin
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaetsklinikum Gießen, Marburg
- Semmelweis Egyetem AOK I.sz. Belgyogyaszati Klinika, Budapest, Hungary
- Italy (3):
  - Presidio Ospedaliero di Castelfranco Veneto, Castelfranco Veneto, Treviso
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Policlinico Umberto I di Roma-Università di Roma La Sapienza, Roma
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Russia (3):
  - FSBI "Kirov SR Institute of Hematology and Blood Transfusion FMBA", Kirov
  - FSBI "Hematological Research Center" MoH of RF, Moscow
  - SBEI HPE "Samara State Medical University" of the MoH of the RF, Samara
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
- United Kingdom (6):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal London Hospital, London, Greater London
  - Royal Free Hospital, London, Greater London
  - St Thomas' Hospital Centre for Haemostasis & Thrombosis, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - University Hospital of Wales, Cardiff, West Glamorgan

REFERENCES:
- [Derived] Tiede A, Allen G, Bauer A, Chowdary P, Collins P, Goldstein B, Jiang HJ, Kӧck K, Takacs I, Timofeeva M, Wolfsegger M, Srivastava S. SHP656, a polysialylated recombinant factor VIII (PSA-rFVIII): First-in-human study evaluating safety, tolerability and pharmacokinetics in patients with severe haemophilia A. Haemophilia. 2020 Jan;26(1):47-55. doi: 10.1111/hae.13878. Epub 2019 Nov 28. PMID 31778283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 study sites in the EU and Russia. 44 participants signed informed consent. Of these, 4 participants were not treated (2 screen failures and 2 participants withdrew from study prior to receiving any dosing).
Pre-assignment Details: 44 participants signed informed consent. Of these, 4 participants were not treated (2 screen failures and 2 participants withdrew from study prior to receiving any dosing).
Groups:
- Cohort 1 - Low Dose: Participants were to receive an infusion of 25±3 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation. Following the washout period, participants were to receive a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
- Cohort 2 - Medium Dose: After data from Cohort 1 have been reviewed and approved by an internal Safety Monitoring Committee, participants were to receive an infusion of 50±5 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation. Following the washout period, participants were to receive a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
- Cohort 3 - High Dose: After data from Cohort 2 have been reviewed and approved by an internal Safety Monitoring Committee, participants were to receive an infusion of 75±5 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation. Following the washout period, participants were to receive a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
Period: Period 1 - ADVATE
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Started | 11 | 16 | 13
Completed | 10 | 15 | 13
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Period: Period 2 - BAX 826
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Started | 10 | 15 | 13
Completed | 10 | 15 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 3 - High Dose: After data from Cohort 2 have been reviewed and approved by an internal Safety Monitoring Committee, participants were to receive an infusion of 75±3 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation. Following the washout period, participants were to receive a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose | Total
Number analyzed (Participants) | 11 | 16 | 13 | 40
Age, Continuous [Median (Full Range); unit: Years] | 34.0 [20 to 59] | 33.0 [19 to 55] | 36.0 [18 to 63] | 34.0 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 11 | 16 | 13 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 10 | 16 | 13 | 39
  Race: Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Serious AEs (SAEs) and Non-serious AEs Occurring After Infusion With BAX 826
Description: Serious Adverse Events and non-serious Adverse Events the occurred after infusion with BAX 826.
Time Frame: Up to 6 weeks ± 4 days post infusion with BAX826.
Population: Participants in Cohort 1, 2 and 3 in Period 2 (receiving BAX 826) are included.
Measure: Number; unit: Adverse Events
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 10 | 15 | 13
Adverse Events
  Any AE | 20 | 12 | 15
  Any AE with outcome = Death | 0 | 0 | 0
  Any serious AE | 0 | 0 | 0
  Any treatment related serious AE | 0 | 0 | 0
  Any moderate or severe serious AE | 0 | 0 | 0
  Any non-serious AE | 20 | 12 | 15
  Any treatment related non-serious AE | 0 | 0 | 0
  Any moderate or severe non-serious AE | 8 | 3 | 4
  Any systemic AE | 1 | 0 | 4
  Any treatment related systemic AE | 0 | 0 | 0
  Any moderate or severe systemic AE | 0 | 0 | 1
  Any local/non-systemic AE | 19 | 12 | 11
  Any treatment related local/non-systemic AE | 0 | 0 | 0
  Any moderate or severe local/non-systemic AE | 8 | 3 | 3
  Any AE leading to study treatment withdrawal | 0 | 0 | 0

2. Primary Outcome: Immediate Tolerability (Vital Signs and Clinical Laboratory Assessments)
Description: Clinically significant results after treatment with investigational product that constitute an AE are counted. Vital signs include body temperature, respiratory rate, pulse rate, and blood pressure. Clinical laboratory results include: Hematology (hemoglobin, hematocrit, red blood cell count, white blood cell count with differential (i.e. basophils, eosinophils, lymphocytes, monocytes and neutrophils), international normalized ratio (INR), mean corpuscular volume (MCV), mean corpuscular hemoglobin concentration (MCHC), platelet count. Clinical Chemistry: sodium, potassium, chloride, bicarbonate, total protein, albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, gamma-glutamyltransferase (GGT), blood urea nitrogen (BUN), creatinine, glucose. Lipid panel: cholesterol, very-low-density lipoprotein (VLDL), low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides
Time Frame: Screening (Day -30 to -2); Advate Administration (Study Day 1) pre & postdose, and Day 4; Advate washout 96 hours to 4 weeks; BAX826 Administration Day 1 pre & postdose, Post BAX826 Day 4, 8, 14, and 23; and study termination visit, week 6 ± 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 13
Participants
  Clinically significant vital signs | 0 | 0 | 0
  Clinically sign. laboratory results after Advate | 0 | 0 | 1
  Clinically sign. laboratory results after BAX826 | 0 | 0 | 3

3. Primary Outcome: Immunogenicity: Inhibitory Antibodies to Factor VIII (FVIII)
Description: Inhibition of FVIII activity by antibodies binding to FVIII were measured using the Nijmegen modification of the Bethesda inhibitor assay.
Time Frame: Screening visit (Day -30 to -2); Advate Administration (Study Day 1) predose; ADVATE wash out period 96 hours to 4 weeks; BAX826 Administration Day 1 predose, and Post BAX826 Day 8; and study termination visit, week 6 ± 4 days
Population: The immunogenicity analysis was performed on the participants of the safety population (participants who received at least one administration of BAX 826 or ADVATE) who have a predose and at least one postdose result.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 10 | 14 | 13
Participants | 0 | 0 | 0

4. Primary Outcome: Immunogenicity: Binding Antibodies to PSA-FVIII (ie BAX 826)
Description: Binding antibodies to PSA FVIII (ie BAX 826) IgG and IgM
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 - Low Dose ADVATE: Participants received an infusion of 25±3 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation.
- Cohort 2 - Medium Dose ADVATE: Participants received an infusion of 50±5 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation.
- Cohort 3 - High Dose ADVATE: Participants received an infusion of 75±3 IU/kg ADVATE followed by a minimum 4-day (96 hours) wash out period including a 3 day PK evaluation.
- Cohort 1 - Low Dose BAX 826: After the 4 day washout period following the infusion of 25±3 IU/kg ADVATE, participants received a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
- Cohort 2 - Medium Dose BAX 826: After the washout period following the infusion of 50±5 IU/kg ADVATE, participants received a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
- Cohort 3 - High Dose BAX 826: After the washout period following the infusion of 75±3 IU/kg ADVATE, participants received a single dose of BAX 826, equivalent to the ADVATE dose they had received, followed by a 7-day PK evaluation.
Arm/Group | Cohort 1 - Low Dose ADVATE | Cohort 2 - Medium Dose ADVATE | Cohort 3 - High Dose ADVATE | Cohort 1 - Low Dose BAX 826 | Cohort 2 - Medium Dose BAX 826 | Cohort 3 - High Dose BAX 826
Number analyzed (Participants) | 10 | 14 | 13 | 10 | 15 | 13
Participants
  IgG: At least 1 positive result (includ.predose) | 1 | 0 | 0 | 1 | 0 | 1
  IgG: Predose negative / Postdose positive | 0 | 0 | 0 | 0 | 0 | 1
  IgM: At least 1 positive result (includ.predose) | 0 | 1 | 0 | 0 | 0 | 1
  IgM: Predose negative / Postdose positive | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Immunogenicity: Binding Antibodies to Factor VIII (FVIII)
Description: Binding antibodies to FVIII IgG and IgM
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose ADVATE | Cohort 2 - Medium Dose ADVATE | Cohort 3 - High Dose ADVATE | Cohort 1 - Low Dose BAX 826 | Cohort 2 - Medium Dose BAX 826 | Cohort 3 - High Dose BAX 826
Number analyzed (Participants) | 11 | 14 | 13 | 10 | 15 | 13
Participants
  IgG: At least 1 positive result (includ.predose) | 0 | 0 | 0 | 1 | 0 | 0
  IgG: Predose negative / Postdose positive | 0 | 0 | 0 | 1 | 0 | 0
  IgM: At least 1 positive result (includ.predose) | 0 | 0 | 0 | 0 | 0 | 0
  IgM: Predose negative / Postdose positive | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Immunogenicity: Anti-polysialic Acid (Anti-PSA) Antibodies
Description: Binding antibodies to PSA (IgG and IgM)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose ADVATE | Cohort 2 - Medium Dose ADVATE | Cohort 3 - High Dose ADVATE | Cohort 1 - Low Dose BAX 826 | Cohort 2 - Medium Dose BAX 826 | Cohort 3 - High Dose BAX 826
Number analyzed (Participants) | 11 | 14 | 13 | 10 | 15 | 13
Participants
  IgG: At least 1 positive result (includ.predose) | 0 | 0 | 0 | 0 | 0 | 0
  IgG: Predose negative / Postdose positive | 0 | 0 | 0 | 0 | 0 | 0
  IgM: At least 1 positive result (includ.predose) | 0 | 1 | 3 | 0 | 1 | 3
  IgM: Predose negative / Postdose positive | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Immunogenicity: Anti-Chinese Hamster Ovary (Anti-CHO) Antibodies
Description: Binding antibodies to CHO
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 10 | 15 | 13
Participants | 0 | 0 | 0

8. Primary Outcome: Immunogenicity: Human Anti-murine Antibodies (HAMA)
Description: Binding antibodies HAMA (IgG)
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 10 | 15 | 13
Participants | 0 | 0 | 0

9. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From 0 to Infinity (AUC0-∞)
Description: Area under the FVIII activity-time curve from zero extrapolated to infinity, calculated by linear-up/log-down trapezoidal method and extrapolated to infinity, calculated as AUC last + C last / lambda z, where Clast is the estimated concentration at the last quantifiable time point
Time Frame: Pre-infusion within 30 minutes; and post-infusion at 15 and 30 minutes, and 1, 3, 6, 9, 12, 24, 32, 48, 56, and 72 hours for both BAX 826 and ADVATE. BAX 826 will also include post-infusion at 96, 120, 144, and 168 hours.
Population: In period 1 (ADVATE) the number of participants is 11,16,12 respectively for Cohorts 1, 2 and 3. In period 2 (BAX 826) the number of participants is 8, 10 and 11 respectively for cohorts 1, 2 and 3 (10 participants were excluded from the PK analysis for period 2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/dL
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
IU*h/dL
  Period 1 (ADVATE) - One Stage Clotting Assay | 901.3 (43.3) | 1771 (30.9) | 2496 (39.3)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 1127 (73.1) | 2363 (24.3) | 2578 (55.0)
  Period 1 (ADVATE) - Chromogenic Assay | 818.9 (38.6) | 1747 (31.0) | 2693 (34.9)
  Period 2 (BAX 826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - Chromogenic Assay | 1234 (67.4) | 2742 (36.4) | 3791 (55.9)

10. Secondary Outcome: Pharmacokinetics: Terminal Half-life (t1/2)
Description: Terminal elimination phase half-life, calculated by (ln2)/lambda z, where lambda z is the terminal rate constant, determined by linear regression of the terminal points of the log-linear FVIII activity-time curve.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
hours
  Period 1 (ADVATE) - One Stage Clotting Assay | 10.57 (39.1) | 11.30 (29.6) | 9.948 (34.8)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 16.18 (41.3) | 16.90 (21.0) | 16.22 (28.1)
  Period 1 (ADVATE) - Chromogenic Assay | 11.23 (35.4) | 11.21 (35.7) | 12.11 (28.5)
  Period 2 (BAX826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX826) - Chromogenic Assay | 16.04 (35.6) | 15.21 (20.2) | 16.72 (28.2)

11. Secondary Outcome: Pharmacokinetics: Mean Residence Time (MRT)
Description: Mean residence time, calculated as (AUMC 0-∞ / AUC 0-∞) - TI / 2, where TI is the time duration of infusion
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
hours
  Period 1 (ADVATE) - One Stage Clotting Assay | 15.55 (39.9) | 16.30 (30.5) | 14.00 (29.7)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 26.96 (43.4) | 28.90 (17.4) | 24.33 (27.8)
  Period 1 (ADVATE) - Chromogenic Assay | 15.23 (36.1) | 14.56 (29.5) | 15.36 (29.1)
  Period 2 (BAX826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX826) - Chromogenic Assay | 24.26 (34.1) | 22.83 (20.3) | 24.10 (28.2)

12. Secondary Outcome: Pharmacokinetics: Total Body Clearance (CL)
Description: Systemic body clearance of drug from plasma, calculated by dose (IU/kg)/AUC0-∞
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: dL/kg*h
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
dL/kg*h
  Period 1 (ADVATE) - One Stage Clotting Assay | 0.02803 (47.0) | 0.02831 (31.4) | 0.02989 (39.3)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 0.02213 (74.8) | 0.02161 (25.4) | 0.02950 (55.8)
  Period 1 (ADVATE) - Chromogenic Assay | 0.03085 (42.2) | 0.02871 (31.5) | 0.02771 (33.7)
  Period 2 (BAX 826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - Chromogenic Assay | 0.02022 (69.4) | 0.01862 (37.4) | 0.02006 (57.0)

13. Secondary Outcome: Pharmacokinetics: Incremental Recovery (IR)
Description: Incremental recovery (IR) at Cmax, calculated as IR = (Cmax - Cpreinfusion) / Dose (IU/kg)
Time Frame: as for outcome 9
Population: In period 1 (ADVATE) the number of participants is 11,15,12 respectively for Cohorts 1, 2 and 3. In period 2 (BAX 826) the number of participants is 8, 10 and 11 respectively for cohorts 1, 2 and 3 (9 participants were excluded from the PK analysis for period 2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU/dL)/(IU/kg)
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 15 | 12
(IU/dL)/(IU/kg)
  Period 1 (ADVATE) - One Stage Clotting Assay | 2.506 (18.1) | 2.594 (17.0) | 3.059 (25.3)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 1.544 (27.5) | 1.560 (22.0) | 1.641 (41.2)
  Period 1 (ADVATE) - Chromogenic Assay | 2.850 (14.6) | 3.194 (13.0) | 3.467 (20.4)
  Period 2 (BAX826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX826) - Chromogenic Assay | 2.391 (26.4) | 2.781 (35.2) | 2.512 (26.2)

14. Secondary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution at steady state is calculated by MRT*CL MRT=Mean residence time CL=Clearance rate
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: dL/kg
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
dL/kg
  Period 1 (ADVATE) - One Stage Clotting Assay | 0.4359 (17.4) | 0.4615 (17.7) | 0.4183 (17.9)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 0.5967 (29.7) | 0.6246 (24.2) | 0.7176 (28.4)
  Period 1 (ADVATE) - Chromogenic Assay | 0.4700 (14.6) | 0.4181 (20.6) | 0.4256 (26.7)
  Period 2 (BAX 826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - Chromogenic Assay | 0.4906 (34.6) | 0.4253 (35.5) | 0.4835 (32.4)

15. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax)
Description: Maximum observed FVIII activity, obtained directly from FVIII activity versus time data
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/dL
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 15 | 12
IU/dL
  Period 1 (ADVATE) - One Stage Clotting Assay | 63.32 (16.4) | 130.06 (16.4) | 228.24 (23.5)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 38.53 (26.7) | 79.65 (21.4) | 124.78 (40.8)
  Period 1 (ADVATE) - Chromogenic Assay | 72.00 (12.8) | 160.16 (12.1) | 258.68 (21.4)
  Period 2 (BAX826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX826) - Chromogenic Assay | 59.65 (23.8) | 142.00 (35.1) | 191.01 (25.7)

16. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration in Plasma (Tmax)
Description: Time of maximum FVIII activity is obtained directly from FVIII activity versus time data
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 15 | 12
hours
  Period 1 (ADVATE) - One Stage Clotting Assay | 0.3000 [0.250 to 1.033] | 0.3330 [0.250 to 1.000] | 0.3170 [0.250 to 3.017]
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 11 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 0.3000 [0.250 to 0.533] | 0.5165 [0.283 to 1.067] | 0.5500 [0.250 to 1.050]
  Period 1 (ADVATE) - Chromogenic Assay | 0.3000 [0.250 to 0.633] | 0.3330 [0.250 to 1.050] | 0.3085 [0.250 to 1.067]
  Period 2 (BAX 826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - Chromogenic Assay | 0.3835 [0.250 to 0.617] | 0.3165 [0.250 to 1.067] | 0.3000 [0.250 to 0.550]

17. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Time Point (AUC0-last)
Description: Area under the FVIII activity-time curve from zero to the last quantifiable FVIII activity, calculated by linear-up/log-down trapezoidal method.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/dL
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
IU*h/dL
  Period 1 (ADVATE) - One Stage Clotting Assay | 861.8 (42.5) | 1712 (30.9) | 2445 (38.3)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 1078 (73.7) | 2296 (25.8) | 2528 (55.9)
  Period 1 (ADVATE) - Chromogenic Assay | 785.4 (39.2) | 1703 (30.3) | 2625 (34.6)
  Period 2 (BAX 826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - Chromogenic Assay | 1181 (70.8) | 2717 (37.4) | 3726 (57.2)

18. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From 0 to 72 Hours (AUC0-72h)
Description: AUC from time zero to exactly 72 hours, calculated by linear-up/log-down trapezoidal method. If the sample at 72 hours is missing, the activity at 72 hours will be interpolated or extrapolated using the last quantifiable activity and the terminal rate constant (lambda z).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/dL
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
IU*h/dL
  Period 1 (ADVATE) - One Stage Clotting Assay | 885.9 (41.8) | 1736 (29.2) | 2463 (37.5)
  Period 2 (BAX 826) - One Stage Clotting Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - One Stage Clotting Assay | 1041 (68.4) | 2168 (23.4) | 2421 (49.7)
  Period 1 (ADVATE) - Chromogenic Assay | 803.3 (37.3) | 1717 (30.0) | 2638 (34.0)
  Period 2 (BAX 826) - Chromogenic Assay: number analyzed (Participants) | 8 | 10 | 11
  Period 2 (BAX 826) - Chromogenic Assay | 1157 (63.5) | 2609 (35.9) | 3556 (51.5)

19. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From 0 to 168 Hours (AUC0-168h) for BAX 826
Description: AUC from time zero to exactly 168 hours, calculated by linear-up/log-down trapezoidal method. If the sample at 168 hours is missing, the activity at 168 hours was interpolated or extrapolated using the last quantifiable activity and the terminal rate constant (lambda z). This parameter will be calculated for BAX 826 only.
Time Frame: Pre-infusion within 30 minutes; and post-infusion at 15 and 30 minutes, and 1, 3, 6, 9, 12, 24, 32, 48, 56, 72, 96, 120, 144, and 168 hours.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/dL
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 8 | 10 | 11
IU*h/dL
  Period 2 (BAX 826) - One Stage Clotting Assay | 1124 (72.9) | 2358 (24.2) | 2572 (54.7)
  Period 2 (BAX 826) - Chromogenic Assay | 1231 (67.2) | 2739 (36.4) | 3783 (55.6)

20. Secondary Outcome: Comparison of Key Pharmacokinetic Parameters by Cohort
Description: The key pharmacokinetic parameters (Area under the concentration-time curve from 0 to infinity (AUC0-∞), Area under the concentration-time curve from 0 to 72 hours (AUC0-72h), Maximum plasma concentration (Cmax), Terminal half-life (t1/2), Mean residence time (MRT) and Total body clearance (CL)) for ADVATE and BAX 826 have been compared.
Time Frame: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Ratio of Geometric Means (%)
Arm/Group | Cohort 1 - Low Dose | Cohort 2 - Medium Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 11 | 16 | 12
Ratio of Geometric Means (%)
  AUC 0-∞: One Stage Clotting Assay | 116.20 [83.53 to 161.64] | 122.53 [108.19 to 138.78] | 100.79 [78.64 to 129.19]
  AUC 0-∞: Chromogenic Assay | 141.10 [98.78 to 201.55] | 155.57 [128.11 to 188.92] | 138.99 [106.10 to 182.08]
  AUC 0-72: One Stage Clotting Assay | 109.28 [80.72 to 147.94] | 115.60 [101.89 to 131.16] | 96.07 [75.91 to 121.58]
  AUC 0-72: Chromogenic Assay | 135.27 [95.99 to 190.63] | 150.69 [124.20 to 182.83] | 133.20 [102.95 to 172.33]
  Cmax: One Stage Clotting Assay | 61.15 [50.43 to 74.15] | 63.28 [57.71 to 69.38] | 54.40 [41.79 to 70.82]
  Cmax: Chromogenic Assay | 82.85 [69.48 to 98.78] | 89.17 [75.31 to 105.58] | 73.68 [60.37 to 89.92]
  t 1/2: One Stage Clotting Assay | 142.10 [115.18 to 175.32] | 147.44 [118.53 to 183.41] | 159.52 [140.28 to 181.40]
  t 1/2: Chromogenic Assay | 136.97 [118.80 to 157.91] | 130.84 [108.73 to 157.45] | 138.28 [124.77 to 153.26]
  MRT: One Stage Clotting Assay | 157.83 [136.90 to 181.95] | 165.99 [146.90 to 187.55] | 171.33 [158.83 to 184.82]
  MRT: Chromogenic Assay | 148.12 [127.70 to 171.82] | 151.69 [136.33 to 168.78] | 156.29 [146.73 to 166.47]
  CL: One Stage Clotting Assay | 85.97 [62.65 to 117.95] | 83.21 [73.83 to 93.78] | 100.98 [77.76 to 131.13]
  CL: Chromogenic Assay | 70.73 [49.67 to 100.72] | 65.44 [54.14 to 79.11] | 73.26 [55.37 to 96.95]

21. Secondary Outcome: Summary of Assessment of Dose Proportionality for BAX 826
Description: Dose Proportionality for BAX 826 was calculated for the parameters Area under the concentration-time curve from 0 to infinity (AUC0-∞), Area under the concentration-time curve from time 0 to the last quantifiable time point (AUC0-last) and Maximum plasma concentration (Cmax).
Time Frame: as for outcome 19
Population: The PK analysis set consists of all subjects that have received at least 1 administration of ADVATE or BAX 826 and are evaluable for PK for one or both treatments.
Measure: Number (95% Confidence Interval); unit: Doubling dose increase
Groups:
- Pharmacokinetic Analysis Data Set: The PK analysis set includes all participants that underwent pharmacokinetic assessments.
Arm/Group | Pharmacokinetic Analysis Data Set
Number analyzed (Participants) | 29
Doubling dose increase
  AUC 0-∞: One Stage Clotting Assay | 1.668 [1.310 to 2.124]
  AUC 0-∞: Chromogenic Assay | 1.979 [1.549 to 2.529]
  AUC 0-last: One Stage Clotting Assay | 1.696 [1.328 to 2.167]
  AUC 0-last: Chromogenic Assay | 2.014 [1.564 to 2.592]
  Cmax: One Stage Clotting Assay | 2.058 [1.772 to 2.389]
  Cmax: Chromogenic Assay | 2.055 [1.782 to 2.369]

ADVERSE EVENTS:
Time Frame: Throughout the study period (total study duration approximately 9 months). For each participant from screening until study termination visit (approximately 6 weeks ± 4 days after BAX 826 administration).
Description: Adverse events were recorded throughout the study from screening to completion/termination visit.
Arm/Group | Cohort 1 - Low Dose ADVATE | Cohort 2 - Medium Dose ADVATE | Cohort 3 - High Dose ADVATE | Cohort 1 - Low Dose BAX 826 | Cohort 2 - Medium Dose BAX 826 | Cohort 3 - High Dose BAX 826
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/16 | 0/13 | 0/10 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/16 | 0/13 | 0/10 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 3/11 | 0/16 | 4/13 | 6/10 | 6/15 | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Low Dose ADVATE (N=11) | Cohort 2 - Medium Dose ADVATE (N=16) | Cohort 3 - High Dose ADVATE (N=13) | Cohort 1 - Low Dose BAX 826 (N=10) | Cohort 2 - Medium Dose BAX 826 (N=15) | Cohort 3 - High Dose BAX 826 (N=13)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 5 | 3 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication. The sponsor requires a review of results communication (e .g. for confidential information) >= 45 days prior to submission and may request an additional delay of <=210 days (e .g. for intellectual property protection).